CLINICAL TRIAL: NCT04548622
Title: Bilateral rTMS Clinical Trial for Persistent Auditory Hallucinations Results for a Terminated Study
Brief Title: Bilateral Repetitive Transcranial Magnetic Stimulation for Auditory Hallucinations Results
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Dr. Ralph Hoffman unexpectedly passed away.
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0409027023_b; R01MH073673-02 (NIH); NARSAD; 2R01MH067073 (NIH)
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Schizophrenia
Keywords: Schizoaffective disorder; Auditory Hallucinations; Voices; Repetitive Transcranial Magnetic Stimulation; rTMS; Wernicke's Area; Middle Temporal Cortex; Persistent Auditory Hallucinations; Previously Participated in "Parent" rTMS Protocol
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hallucinations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Non-randomized bilateral rTMS (Experimental): Active bilateral rTMS to left/right Wernicke's area and opposite side middle temporal gyrus
  Interventions: Device: Magstim Rapid 2 system triggering Magstim Super Rapid system

INTERVENTIONS:
Device: Magstim Rapid 2 system triggering Magstim Super Rapid system — Week 1 treatment includes rTMS for 5 sessions to both the left and right Wernicke's area (BA22) synchronous with rTMS to opposite hemisphere middle temporal cortex (BA21). Week 2 treatment includes rTMS given for 5 sessions with positions reversed (e.g., if Wernicke's stimulation was on the left during Week 1, position of rTMS will switch to the right side during Week 2 and vice-versa). As in Week 1, active rTMS will also be given synchronously to the opposite hemisphere middle temporal cortex. Weeks 3 and 4 include 10 stimulation sessions to the configuration of sites producing greater improvement in comparing results of Week 1 and Week 2. rTMS for each stimulation session will be given at 1-Hertz (once per second) for 16 minutes without interruption.

SUMMARY:
The primary purpose of this study was to conduct fMRI neuroimaging studies prior to and subsequent to the rTMS intervention. The intent was to ascertain changes in regional brain activation and connectivity that most robustly predict level of improvement in auditory hallucinations elicited by bilateral rTMS as assessed by the primary outcome variables.

DETAILED DESCRIPTION:
This study is an extension of previous clinical trials (NCT00308997 and NCT00567281) that were initiated in 2006. This study record provides the results for the amended study NCT00567281 (originally called a 'third arm') that was discontinued following the passing of Dr. Ralph Hoffman. The primary purpose of the study was to conduct fMRI neuroimaging studies prior to and subsequent to the rTMS intervention. The intent was to ascertain changes in regional brain activation and connectivity that most robustly predict level of improvement in auditory hallucinations elicited by bilateral rTMS as assessed by our primary outcome variables. It was hoped that this combined fMRI/rTMS study would provide critical new insights into the neurobiological basis of auditory hallucinations.

The results presented are what was summarized following Dr. Hoffman's passing and were compiled by Dr. Philip Corlett.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in our "parent" rTMS trial with passage of at least six months since last received active rTMS

Exclusion Criteria:

* Active substance abuse or alcohol abuse
* Pregnancy
* Dose or type of psychiatric medication changed within the 4 weeks prior to study entry
* Recent head trauma, seizures, or significant unstable medical condition

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Corlett, PhD, Principal Investigator — Yale University Department of Psychiatry
Locations (1):
- Department of Psychiatry, Yale School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Background] Hoffman RE, Gueorguieva R, Hawkins KA, Varanko M, Boutros NN, Wu YT, Carroll K, Krystal JH. Temporoparietal transcranial magnetic stimulation for auditory hallucinations: safety, efficacy and moderators in a fifty patient sample. Biol Psychiatry. 2005 Jul 15;58(2):97-104. doi: 10.1016/j.biopsych.2005.03.041. PMID 15936729
- [Background] Hoffman RE, Boutros NN, Hu S, Berman RM, Krystal JH, Charney DS. Transcranial magnetic stimulation and auditory hallucinations in schizophrenia. Lancet. 2000 Mar 25;355(9209):1073-5. doi: 10.1016/S0140-6736(00)02043-2. PMID 10744097
- [Background] Hoffman RE, Hampson M, Wu K, Anderson AW, Gore JC, Buchanan RJ, Constable RT, Hawkins KA, Sahay N, Krystal JH. Probing the pathophysiology of auditory/verbal hallucinations by combining functional magnetic resonance imaging and transcranial magnetic stimulation. Cereb Cortex. 2007 Nov;17(11):2733-43. doi: 10.1093/cercor/bhl183. Epub 2007 Feb 13. PMID 17298962
- [Background] Hoffman RE, Anderson AW, Varanko M, Gore JC, Hampson M. Time course of regional brain activation associated with onset of auditory/verbal hallucinations. Br J Psychiatry. 2008 Nov;193(5):424-5. doi: 10.1192/bjp.bp.107.040501. PMID 18978327
- See also: Click here for a description of rTMS trials of auditory hallucinations at Yale — http://www.med.yale.edu/psych/clinics/rTMS.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-randomized Bilateral rTMS
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Non-randomized Bilateral rTMS
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: PANSS Composite Positive Symptoms Hallucination Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia.The PANSS positive symptoms hallucinication score has a range of 1-7. Higher scores indicate more severe positive symptoms in patients with schizophrenia.
Time Frame: baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-randomized Bilateral rTMS
Number analyzed (Participants) | 15
units on a scale
  Baseline | 5.19 (0.85)
  4 weeks | 4.19 (1.07)
Statistical Analysis 1: Comparison: Non-randomized Bilateral rTMS; Test type: Superiority; p = 0.01, t-test, 2 sided

2. Primary Outcome: PANSS Composite Negative Symptom Scale
Description: The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia.The PANSS negative scale has 7 Items, with a minimum score of 7 and a maximum score of 49. Higher scores indicate more severe negative symptoms in patients with schizophrenia.
Time Frame: baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-randomized Bilateral rTMS
Number analyzed (Participants) | 15
units on a scale
  Baseline | 16.9 (5.22)
  4 weeks | 12.53 (4.54)
Statistical Analysis 1: Comparison: Non-randomized Bilateral rTMS; Test type: Superiority; p = 0.004, t-test, 2 sided

3. Primary Outcome: PANSS Total Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia.The PANSS total score has a minimum score of 30 and a maximum score of 210. Higher scores indicate more severe symptoms in patients with schizophrenia.
Time Frame: baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-randomized Bilateral rTMS
Number analyzed (Participants) | 15
units on a scale
  Baseline | 67.8 (17.9)
  4 weeks | 53.2 (14.9)
Statistical Analysis 1: Comparison: Non-randomized Bilateral rTMS; Test type: Superiority; p = 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Arm/Group | Non-randomized Bilateral rTMS
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes